CLINICAL TRIAL: NCT06639750
Title: Dynamic Evaluation of Composition and Evolution of Respiratory Viroma/Microbioma of Patients Who Have Undergone Hematopoiteic Stem Cell Transplantation (HSCT), as a Possible Biomarker of Occurrence of Post-HSCT Pulmonary Complications.
Brief Title: Respiratory Microbioma and Respiratory Complications After Hematopoietic Stem Cell Transplantion
Acronym: VIREMIG
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: VIREMID 24-0157
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Hematopoietic Stem Cell Transplantation; Microbioata; Respiratory Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Blood sample and nasal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Allogeneic haematopoietic stem cell transplantation (AHSCT) is a therapeutic resource for many haemopathies. The number of HSCTs has risen sharply in recent years due to the use of attenuated conditioning, which has increased the risk of non-haematological complications. Pulmonary pathologies are a frequent cause of complications following HSCA, both infectious and non-infectious(1,3,4).

Among these, late non-infectious pulmonary complications (LNIPC), all taken together, occur in 25% of post-HSCA cases(1). These NIPCs, the most common of which is bronchiolitis obliterans, significantly alter the prognosis(4,5). The pathophysiology of CPTNI is poorly understood, but it seems that the occurrence of a viral respiratory infection (pre- or post-ACSH) may be a potential trigger for the onset of CPTNI(1). These viral infections can become "chronic", given that viral clearance is impaired by the underlying immunodepression, and can thus cause chronic inflammation leading to the fibrosing and irreversible process of obliterative bronchiolitis(6). Given the prognostic importance of this type of CPTNI, it seems essential to gain a better understanding of its pathophysiology, which may involve a number of mechanisms: cellular expression of the graft and its evolution, disruption of the host response (innate immunity) following viral infection, influence of the microbiome and alteration of epithelial repair(1,3,5). Interest in the digestive and respiratory microbiome has been growing in recent years(7-9). The literature is gradually being enriched with data on the links between infection, the microbiome and chronic respiratory pathology and, in the post-HSCA context, a potential link between the enteric microbiome and Chronic Graft Versus Host Disease (cGVHD).

A pilot study comparing respiratory microbiomes using sequencing and metatranscriptomic analysis on 20 respiratory samples (nasopharyngeal swab and bronchoalveolar lavage pairs) taken under the conditions of the proposed study showed that the technique was highly feasible and highly sensitive.

The aim of this study is therefore to use meta-genomics to investigate the respiratory virome/microbiome in a population of patients who have undergone HSCA: eukaryotic and prokaryotic viruses, bacterial expression and the expression (meta-transcriptomics) of graft-derived cell lines and their possible association with the occurrence of post-HSCA respiratory complications (infectious and non-infectious).

No study has assessed the link between the composition of the respiratory virome/microbiome and the occurrence of respiratory events (infectious and CPTNI post ACSH), but also more broadly the link with the composition of the microbiome in the broad sense (respiratory virome, respiratory and digestive microbiota).

The aim of this study is to establish a respiratory viral and bacterial map as a possible biomarker of the occurrence of respiratory events (infectious and CPTNI), thus enabling more personalised monitoring of patients at risk of CPTNI and management of immunosuppressive treatment of patients at risk of an infectious episode, with risk assessment based on the composition of the respiratory virome.

The interest of this study is that it is multidisciplinary and transdisciplinary, studying the respiratory pathologies and infections of haematology patients and combining clinical and fundamental research, with expected spin-offs for direct patient care (personalised monitoring and management of immunosuppressive treatments).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 or over
* French-speaking
* Followed in the centre's haematology department with a project for a haematopoietic stem cell allograft
* Whatever the haemopathy, previous treatments, type of transplant (pheno, geno, haplo-identical), type of graft (bone marrow, peripheral stem cells, cord blood), any conditioning (myeloablative or non-myeloablative), any immunosuppressive protocol.
* Be affiliated to the social security system
* Person able to understand the information and sign the consent form.
* Informed consent must be collected and signed

Exclusion Criteria:

* Refusal to take part in the research
* Failure to sign the consent form
* Contraindication to nasopharyngeal swabbing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients receiving an allogeneic hematopoietic stem cell transplant, whatever the underlying pathology.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
respiratory complications | From enrollment to the end of follow up at 2 years after HSCT